CLINICAL TRIAL: NCT03450889
Title: Effectiveness of a Personalized Endoscopic Surveillance Protocol for Patients With Serrated Polyposis Syndrome
Brief Title: Personalized Surveillance Protocol for Serrated Polyposis Syndrome
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: CA659011
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Serrated Polyposis Syndrome; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention arm: This study uses only one arm. All patients in this intervention arm will be surveyed using the aforementioned study protocol, which means patients will undergo a colonoscopy (or sigmoidoscopy in patients with previous subtotal colectomy) with surveillance intervals of either 1 or 2 years, depending on the amount and type of polyps resected during previous surveillance.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — Patients will undergo surveillance colonoscopies, with intervals of 1 or 2 years depending on the amount and type of polyps resected during last colonoscopy.
  In case patients underwent subtotal colectomy, the term 'colonoscopy' should be replaced with 'sigmoidoscopy'.

SUMMARY:
Serrated polyposis syndrome (SPS) is a condition characterized by the presence of multiple serrated polyps (SPs) spread throughout the colorectum and is associated with an increased risk of colorectal cancer (CRC). SPS is defined by the World Health Organization (WHO) as the presence of at least 5 SPs proximal to the sigmoid colon, of which 2 ≥10 mm in size (WHO criterion 1), the presence of at least 1 SP proximal to the sigmoid and a first degree relative with SPS (WHO criterion 2), or more than 20 SPs spread throughout the colon (WHO-criterion-3). In practice only WHO 1 and WHO 3 criteria are used.

The condition seems rather common and more prevalent than other polyposis syndromes such as familial adenomatous polyposis (FAP) (1:13.000).

Several retrospective studies have shown that patients with SPS have an increased risk of developing CRC during endoscopic surveillance. Close endoscopic surveillance to prevent malignant progression of polyps has therefore been advised by several expert groups. However, due to a shortage of prospective data the optimal treatment and surveillance approach is largely unknown.

The current study aims to prospectively evaluate the effectiveness and feasibility of a personalized surveillance protocol for patients with SPS to prevent CRC that is being used in several Dutch and Spanish hospitals. Furthermore, the polyp burden, colonoscopy complication risk and rate of conversion from endoscopic surveillance to colorectal surgery will be examined.

For this purpose, all eligible SPS patients are prospectively enrolled 2013 onwards, and surveyed according to the study protocol. Based on the amount and characteristics of the polyps encountered during surveillance colonoscopy, the next colonoscopy will be scheduled after either 1 year or 2 years.

Patients will undergo surveillance after 1 year in case of:

* Advanced adenoma (≥ 10 mm and/or high-grade dysplasia and/or 25% villous component)
* Serrated polyp ≥ 10mm and/or SP containing dysplasia
* Cumulative ≥5 sessile serrated polyps (SSPs) (irrespective of size), adenomas (irrespective of size) and/or hyperplastic polyps (HPs) ≥5mm
* Surgery needed during previous (clearing or surveillance) endoscopy

Patients will undergo surveillance after 2 years in case none of above is reached

DETAILED DESCRIPTION:
This study has an international multi-centre prospective cohort design. The study will be directed by the Academic Medical Centre (AMC), Amsterdam, the Netherlands.

Population base All patients treated at one of the participating centres will be eligible for this study.

Protocol violations Incomplete endoscopic excision of polyps without proper re-colonoscopy Prolonged interval within surveillance colonoscopies (Exceeding protocol with >1 year)

Sample size calculation No sample size calculation is performed, because of the observational design of this study. All eligible patients will be included, unless an exclusion criterion is met. The envisioned number of patients to be included is around 500.

Institutional review board This study is conducted in accordance with the research code of our Institutional Review Board (IRB) on human experimentation as well as in agreement with the Helsinki Declaration. The IRB decided that the study did not apply to the requirements of the Medical Research Involving Human Subjects Act (WMO), as data were collected during routine care and no additional patient interventions will be undertaken. Therefore also no informed consent is needed for this study. The study protocol will be registered on a publicly accessible website register.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SPS WHO 1 criterion (cumulative ≥ 5 histologically diagnosed SPs proximal to the sigmoid colon, of which 2 ≥ 10mm in diameter) and/or WHO 3 criterion (cumulative ≥ 20 SPs spread throughout the colon, at least 3 of the SPs will have to be situated proximal to the sigmoid colon).
* Age 18 years or older

Exclusion Criteria:

* - Germline mutation for hereditary colorectal cancer syndrome (e.g. familial adenomatous polyposis, Lynch syndrome. Not including heterozygous MUTYH mutation)
* Inflammatory bowel disease
* Proctocolectomy
* History of radiotherapy in abdominal region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated at one of the participating centres during the study will be eligible for this study if they fulfill the inclusion criteria.
  Patients will only be included in the final analyses if they underwent at least one protocolled surveillance coloscopy after complete clearing.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of colorectal cancer during protocolled endoscopic surveillance | Up to five years
  Incidence of colorectal cancer after complete clearing of all relevant polyps, during protocolled surveillance phase.

SECONDARY OUTCOMES:
Incidence of advanced neoplasia during protocolled surveillance phase | Up to five years
  Advanced neoplasia is defined as: (tubulo)villous adenomas, adenomas with high-grade dysplasia or diameter of at least 10mm; serrated polyp with dysplasia, traditional serrated adenomas or serrated polyps with a diameter of at least 10mm.
  CRC is not included in this definition, since CRC is the primary outcome measure in this study.
Incidence of non-advanced relevant neoplasia during protocolled surveillance phase | Up to five years
  Non-advanced relevant neoplasia is defined as tubular adenomas <10mm, sessile serrated lesions <10mm, hyperplastic polyps of 5-9mm.
the ratio of annual and biennial surveillance advise | Up to five years
  Patients will undergo surveillance colonoscopies with intervals of 1 or 2 years. This outcome measure expresses the relative frequency of these surveillance intervals.
Incidence of conversion to preventive colorectal surgery | Up to five years
  How often is preventive colorectal surgery needed during surveillance, for example because of unresectable polyps. This does not include colorectal surgery due to colorectal cancer.
Incidence of post-colonoscopy complications | Up to five years
  Incidence of complications after colonoscopy (this does not include complications that are effectively solved during the procedure). Severity expressed using Clavien Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided